CLINICAL TRIAL: NCT01057745
Title: Ovarian Tissue Freezing Prior to Chemotherapy or Radiation Therapy: a Study by the Oncofertility Consortium
Brief Title: Ovarian Freezing Before Cancer Treatment
Status: Terminated | Type: Observational
Why Stopped: This treatment is now considered standard of care
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 806062
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Effects of Chemotherapy
Keywords: woman; chemotherapy; radiation; fertility preservation; cryobank

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ovarian tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Women of reproductive age who will undergo cancer treatment may participate in a study to surgically remove ovarian tissue and store it, frozen, for their potential use in the future. 20% of collected tissue will be used for research.

DETAILED DESCRIPTION:
Chemotherapy and radiation therapy for cancer can compromise the ability to become pregnant. Experiments in animals and humans have tried to collect, freeze and store eggs to see if they can be saved for possible later use. While studies are promising, it is still uncertain whether such approaches will ultimately prove to be useful in practice for achieving pregnancy in humans. The main purpose of this study is to see whether it is possible to remove and store ovarian tissues by freezing. It is hoped that, in the future, frozen, stored ovarian tissue can be used to achieve pregnancy. Before receiving chemotherapy or radiation therapy, subjects will have a piece of the ovaries, or one of two ovaries, removed by surgery. The tissues will be frozen by a special method in an effort to prevent the eggs from being damaged. The majority (80%) of the tissue will be stored for potential use in case the patient is unable to achieve pregnancy in the future, and part of the tissue (20%) will be used for studying how the eggs can be grown in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Female patient between the ages of 18 and 42 years.
* In need of imminent cancer treatment, including surgery, chemotherapy or radiation therapy, which is viewed as likely to result in a permanent and complete loss of subsequent ovarian function or have a health condition that will result in premature ovarian failure. These include, but are not limited to: abdominopelvic irradiation, total body irradiation, alkylating-intensive chemotherapy, and removal of ovaries as part of their cancer treatment.
* Reasonably good health.
* Two ovaries.
* Able to defer definitive cancer therapy for approximately 3 days until the patient recovers from laparoscopic oophorectomy.

Exclusion Criteria:

* Patients considered as high risk for surgical complications will be excluded from the research protocol.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2007-06-12 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Follicular development in vitro | 5 years
  Several factors, including 3-dimensional biogel scaffolds,growth factors, hormones and other culture conditions, will be investigated as they relate to successful maturation of immature follicles obtained from ovarian tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa Gracia, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Fertility Care, 3701 Market Street, Suite 800, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Gracia CR, Chang J, Kondapalli L, Prewitt M, Carlson CA, Mattei P, Jeffers S, Ginsberg JP. Ovarian tissue cryopreservation for fertility preservation in cancer patients: successful establishment and feasibility of a multidisciplinary collaboration. J Assist Reprod Genet. 2012 Jun;29(6):495-502. doi: 10.1007/s10815-012-9753-7. Epub 2012 Apr 1. PMID 22466745